CLINICAL TRIAL: NCT06670209
Title: A Phase I, Open-label, Fixed-sequence Study to Evaluate the Effect of Repeated Subcutaneous Injections of GZR18 Injection on the Pharmacokinetics of Oral Metformin Hydrochloride Tablets in Overweight/Obese Subjects
Brief Title: A Phase I Clinical Study to Evaluate the Effect of GZR18 Injection on the Pharmacokinetics of Oral Metformin Hydrochloride Tablets in Overweight/Obese Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GZR18-T2D-103
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Drug: GZR18 and metformin

INTERVENTIONS:
Drug: GZR18 and metformin — GZR18: 3 mg-18 mg Metformin: 500 mg

SUMMARY:
This is a single-center, open-label, fixed-sequence phase I clinical study to evaluate the effect of multiple subcutaneous injections of GZR18 Injection on the pharmacokinetics of multiple oral doses of metformin hydrochloride tablets.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese Chinese subjects, who voluntarily sign the Informed Consent Form (ICF), can receive subcutaneous injection, fully understand the content, process and possible adverse reactions of the trial, and are able to follow the regulations on contraindications and restrictions specified in this protocol.
* Male or female, 18 to 50 years of age at signing the ICF (both inclusive).
* Weight ≥ 50 kg and body mass index (BMI) within 24-33 kg/m2 (both ends inclusive) at screening.
* Subjects of childbearing potential with no birth plan from the signing of ICF to 3 months after the last dose, willingness to take effective contraceptive measures, and no plan for sperm or ovum donation. Females of childbearing potential must not be lactating and must have negative results of pregnancy tests at screening and Visit 2 (prior to enrollment).

Exclusion Criteria:

* Subjects with a previous or existing history of heart, liver, kidney, gastrointestinal tract, respiratory system, nervous system, psychiatric disease, malignant tumor and other diseases that are judged by the investigator to have an impact on pharmacokinetics and safety evaluation.
* History or existing diseases that increase the risk of subjects, such as hypoglycaemia, acute or chronic pancreatitis, pancreatic injury, history of symptomatic gallbladder disease; cholelithiasis with high risk of acute biliary pancreatitis at screening (e.g., silt-like lithiasis, gallbladder ≤ 5 mm in diameter and bile duct stone, etc.).
* Subjects with previous or existing diseases that significantly affect drug absorption, metabolism or excretion, such as history of active peptic ulcer or haemorrhage, inflammatory bowel disease, abnormal gastric emptying (such as gastric paresis or pyloric stenosis, gastric outlet obstruction), long-term use (continuous for ≥ 1 week) of drugs that affect gastrointestinal motility (including but not limited to domperidone, mosapride, macrolides).
* Subjects with severe infection or unexplained infection within 4 weeks before screening.
* Major surgery within 6 months prior to screening, or scheduled surgery or hospitalization during the study.
* History of drug abuse prior to screening; or positive results for drug abuse at screening.
* Subjects who used nicotine-containing products within 3 months prior to screening or are screened positive for nicotine in urine.
* Other factors that make subjects unqualified to participate in this trial as judged by the Investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-03-19 (Estimated); Study Completion 2025-03-19 (Estimated)

PRIMARY OUTCOMES:
Cmax,ss | 24 hours
AUC0-tau | 24 hours